CLINICAL TRIAL: NCT04279314
Title: A 40-Week, Open-label Extension Study of Trofinetide for the Treatment of Girls and Women With Rett Syndrome
Brief Title: Open-Label Extension Study of Trofinetide for the Treatment of Girls and Women With Rett Syndrome
Acronym: LILAC™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-2566-004
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Results first posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — trofinetide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Trofinetide (Experimental)
  Interventions: Drug: Trofinetide

INTERVENTIONS:
Drug: Trofinetide — Trofinetide solution of 30-60 mL based on subject's weight at Baseline, administered twice daily by mouth or gastrostomy tube (G-tube)

SUMMARY:
To investigate the safety and tolerability of long-term treatment with oral trofinetide in girls and women with Rett syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Has completed the Week 12/End-of-treatment visit of the antecedent study, Study ACP-2566-003
2. Met all entry criteria for the antecedent study
3. May benefit from long-term treatment with open-label trofinetide in the judgment of the Investigator
4. Can still swallow the study medication provided as a liquid solution or can take it by gastrostomy tube
5. The subject's caregiver is English-speaking and has sufficient language skills to complete the caregiver assessments
6. Subject and caregiver(s) must reside at a location to which study drug can be delivered and have been at their present residence for at least 3 months prior to Baseline

Exclusion Criteria:

1. Began treatment with growth hormone during the antecedent study
2. Began treatment with IGF-1 during the antecedent study
3. Began treatment with insulin during the antecedent study
4. Has developed a clinically significant cardiovascular, endocrine (such as hypo- or hyperthyroidism, Type 1 diabetes mellitus, or uncontrolled Type 2 diabetes mellitus), renal, hepatic, respiratory, or gastrointestinal disease (such as celiac disease or inflammatory bowel disease) or has major surgery planned during the study
5. Subject is judged by the Investigator or the Medical Monitor to be inappropriate for the study due to AEs, medical condition, or noncompliance with investigational product or study procedures in the antecedent study
6. Has a clinically significant abnormality in vital signs at Baseline
7. Has a QTcF interval of >450 ms on the Baseline ECG performed before the first dose of trofinetide is given in the present study
8. Has developed a clinically significant ECG finding during the antecedent study

Additional inclusion/exclusion criteria apply. Patients will be evaluated at baseline to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically, if it is determined that their baseline health and condition do not meet all prespecified entry criteria).

Ages: 5 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 154 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Translational Genomics Research Institute (TGen), Phoenix, Arizona
  - University of California, San Diego, La Jolla, California
  - UC Davis MIND Institute, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children Medical Services, Tampa, Florida
  - Emory Genetics Clinical Trial Center, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Kennedy Krieger Institute - Clinical Trials Unit, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Washington University School of Medicine, St. Louis Children's Hospital, St Louis, Missouri
  - Montefiore Medical Center, Children's Hospital at Montefiore, The Bronx, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Percy AK, Neul JL, Benke TA, Berry-Kravis EM, Glaze DG, Marsh ED, An D, Bishop KM, Youakim JM. Trofinetide for the treatment of Rett syndrome: Results from the open-label extension LILAC study. Med. 2024 Sep 13;5(9):1178-1189.e3. doi: 10.1016/j.medj.2024.05.018. Epub 2024 Jun 24. PMID 38917793
- [Derived] Parent H, Ferranti A, Niswender C. Trofinetide: a pioneering treatment for Rett syndrome. Trends Pharmacol Sci. 2023 Oct;44(10):740-741. doi: 10.1016/j.tips.2023.06.008. Epub 2023 Jul 16. PMID 37460385

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trofinetide
Started | 154
Completed | 84
Not Completed | 70
Not completed — Adverse Event | 55
Not completed — Withdrawal by Subject | 5
Not completed — Lack of Efficacy | 5
Not completed — Protocol Violation | 3
Not completed — Other (not COVID-19 related) | 2

BASELINE CHARACTERISTICS:
Groups:
- Trofinetide: All subjects enrolled and treated with trofinetide
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.0 (4.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 143
  More than one race | 0
  Unknown or Not Reported | 4
Height [Mean (Standard Deviation); unit: cm] | 128.60 (1.229)
Weight [Mean (Standard Deviation); unit: kg] | 29.28 (0.869)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 17.03 (0.285)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Treatment-emergent Adverse Events (TEAEs), Percentage of Subjects With Serious Adverse Events (SAEs), and Percentage of Subjects With Withdrawals Due to AEs
Description: Percentage of subjects with treatment-emergent adverse events (TEAEs), percentage of subjects with serious adverse events (SAEs), and percentage of subjects with withdrawals due to AEs
Time Frame: 40 Weeks Treatment Duration
Measure: Count of Participants; unit: Participants
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
Participants
  Percentage of subjects with TEAEs | 132
  percentage of subjects with SAEs | 19
  Percentage of subjects withdrawals due to AEs | 48

2. Primary Outcome: Subjects (N, %) With Post-baseline Potentially Clinically Important Changes in ECG
Description: Potentially clinically important ECG changes were defined in the study protocol as absolute QTcF interval >500 ms or QTcF interval change from the baseline value of previous study ACP-2566-003 of >60 ms
Time Frame: 40 Weeks Treatment Duration
Measure: Count of Participants; unit: Participants
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
Participants | 2

3. Primary Outcome: Subjects (N, %) With Post-baseline Potentially Clinically Important Changes in Vital Signs
Description: Potentially clinically important changes in vital signs were defined in the study protocol as:
  systolic blood pressure (SBP) ≥180 mmHg and increased ≥20 mmHg from baseline; SBP ≤90 mmHg and decreased ≥20 mmHg from baseline; diastolic blood pressure (DBP) ≥ 105 mmHg and increased ≥15 mmHg from baseline; DBP ≤50 mmHg and decreased ≥15 mmHg from baseline; Pulse ≥120 bpm and increased ≥15 bpm from baseline; Pulse ≤50 bpm and decreased ≥15 bpm from baseline
Time Frame: 40 Weeks Treatment Duration
Measure: Count of Participants; unit: Participants
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
Participants
  SBP ≥180 mmHg and increased ≥20 mmHg from baseline | 0
  SBP ≤90 mmHg and decreased ≥20 mmHg from baseline | 11
  DBP ≥ 105 mmHg and increased ≥15 mmHg from baseline | 0
  DBP ≤50 mmHg and decreased ≥15 mmHg from baseline | 13
  Pulse ≥120 bpm and increased ≥15 bpm from baseline | 14
  Pulse ≤50 bpm and decreased ≥15 bpm from baseline | 0

4. Primary Outcome: Subjects (N, %) With Post-baseline Potentially Clinically Important Changes in Body Weight
Description: Potentially clinically important changes in body weight were defined in the study protocol as:
  Weight increase ≥7% from baseline; Weight decrease ≥7% from baseline
Time Frame: 40 Weeks Treatment Duration
Measure: Count of Participants; unit: Participants
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
Participants
  Weight increase ≥7% from baseline | 44
  Weight decrease ≥7% from baseline | 20

5. Primary Outcome: Subjects (N, %) With Post-baseline Potentially Clinically Important Changes
Description: Potentially clinically important changes in laboratory parameters were defined in the study protocol as:
  Sodium ≤125 mmol/L; Sodium ≥155 mmol/L; Potassium ≤3.0 mmol/L; Potassium ≥5.5 mmol/L; Chloride ≤85 mmol/L; Chloride ≥120 mmol/L; Calcium <2.0 mmol/L; Calcium >2.0 mmol/L; Blood urea nitrogen ≥10.71 mmol/L; Creatinine >1.5 x upper limit of normal (ULN); Uric acid ≥505.75 μmol/L; Lactate dehydrogenase ≥3 x ULN; Glucose ≤2.48 mmol/L; Glucose ≥11 mmol/L; Albumin ≤26 g/L; Albumin ≥60 g/L; Protein ≤50 g/L; Protein ≥100 g/L; Alanine aminotransferase ≥3 x ULN; Aspartate aminotransferase ≥3 x ULN; Gamma glutamyl transpeptidase ≥3 x ULN; Alkaline phosphatase ≥3 x ULN; Bilirubin ≥1.5 x ULN
Time Frame: 40 Weeks Treatment Duration
Population: Subjects with at least 1 post-baseline value for the given parameter (n=151 for all parameters, except LDH (n=150) and AST (=150)
Measure: Count of Participants; unit: Participants
Arm/Group | Trofinetide
Number analyzed (Participants) | 151
Participants
  Sodium ≤125 mmol/L | 0
  Sodium ≥155 mmol/L | 1
  Potassium ≤3.0 mmol/L | 0
  Potassium ≥5.5 mmol/L | 0
  Chloride ≤85 mmol/L | 0
  Chloride ≥120 mmol/L | 1
  Calcium <2.0 mmol/L | 0
  Calcium >2.0 mmol/L | 0
  BUN ≥10.71 mmol/L | 0
  Creatinine >1.5 x ULN | 0
  Uric acid ≥505.75 μmol/L | 0
  Lactate dehydrogenase ≥3× ULN | 0
  Glucose ≤2.48 mmol/L | 4
  Glucose ≥11 mmol/L | 1
  Albumin ≤26 g/L | 2
  Albumin ≥60 g/L | 0
  Protein ≤50 g/L | 1
  Protein ≥100 g/L | 0
  ALT ≥3× ULN | 14
  AST ≥3× ULN | 0
  GGT ≥3× ULN | 4
  ALP ≥3× ULN | 0
  Bilirubin ≥1.5× ULN | 0

6. Secondary Outcome: Rett Syndrome Behaviour Questionnaire (RSBQ) Total Score Change From Baseline to Week 40
Description: The RSBQ is a 45-item caregiver-completed rating scalescale includes 45 items, 39 of them grouped into 8 subscales, whose ratings reflect the severity and frequency of symptoms. Items are rated as 0 (not true), 1 (somewhat or sometimes true), or 2 (very true). The 8 subscales are general mood, breathing problems, hand behavior, face movements, body rocking/expressionless face, night-time behaviors, fear/anxiety, and walking/standing. Scores for item 31 are reversed in the calculation of the total score. The total score ranges from 0 to 90 and is calculated as the sum of the item scores. Higher scores mean worse behaviour.
Time Frame: 40 Weeks Treatment Duration
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
score on a scale | -2.9 (1.17)

7. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score at Week 40
Description: To rate how much the subject's illness has improved or worsened relative to a baseline state, a 7-point scale is used from 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse. Higher CGI-I scores denote more severe illness and less improvement in the illness.
Time Frame: 40 Weeks Treatment Duration
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Placebo/Trofinetide: Subject received placebo in the parent study and trofinetide in the current study
- Trofinetide/Trofinetide: Subject received trofinetidein the parent study and trofinetide in the current study
Arm/Group | Placebo/Trofinetide | Trofinetide/Trofinetide
Number analyzed (Participants) | 85 | 69
score on a scale | 3.2 (0.14) | 3.1 (0.11)

8. Secondary Outcome: Communication and Symbolic Behavior Scales Developmental Profile™ Infant-Toddler Checklist - Social Composite Score (CSBS-DP-IT Social) Change From Baseline to Week 40
Description: Scale to assess communication and pre-linguistic skills in children 12-24 months (or older children with developmental delay). The Checklist consists of 24 questions ranging from 0 to 4 points within each of 7 Clusters. 0 points are given for"Not Yet", 1 point for "Sometimes", or 2 points for "Often". For items describing a series of numbers or ranges, 0 points are given for "None" and 1 to 4 points for items containing numbered choices.
  The Social Composite score is one of 3 composite scores. It comprises 13 items in skill areas "Emotion and Eye Gaze" (items 1 to 4), "Communication" (items 5 to 8), and "Gestures" (items 9 to 13). The Social Composite raw score (items 1 to 13), ranging from 0 to 26, is calculated as the sum of the item scores. Higher Social Composite raw scores indicate better social communication development.
Time Frame: 40 Weeks Treatment Duration
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
score on a scale | 0.5 (0.26)

9. Secondary Outcome: Overall Quality of Life Rating of the Impact of Childhood Neurologic Disability Scale (ICND) Change From Baseline to Week 40
Description: The overall quality of life score rating of the ICND ranges from 1 ("Poor") to 6 ("Excellent"); lower overall quality of life scores indicate lower quality of life.
Time Frame: 40 Weeks Treatment Duration
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
score on a scale | 0.2 (0.09)

10. Secondary Outcome: Rett Syndrome Clinician Rating of Hand Function (RTT-HF) Change From Baseline to Week 40
Description: The RTT-HF is a clinician completed clinical assessment of the subject's ability to use her hands for functional purposes. The assessment is made on an 8-point Likert scale (0-7) with 0 denoting normal functioning and 7 the most severe impairment
Time Frame: 40 Weeks Treatment Duration
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
score on a scale | -0.1 (0.09)

11. Secondary Outcome: Rett Syndrome Clinician Rating of Ambulation and Gross Motor Skills (RTT-AMB) Change From Baseline to Week 40
Description: The RTT-AMB is a clinician completed clinical assessment of the subject's ability to sit, stand, and ambulate. The assessment is made on an 8-point Likert scale (0-7) with 0 denoting normal functioning and 7 the most severe impairment.
Time Frame: 40 Weeks Treatment Duration
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
score on a scale | -0.2 (0.09)

12. Secondary Outcome: Rett Syndrome Clinician Rating of Ability to Communicate Choices (RTT-COMC) Change From Baseline to Week 40
Description: The RTT-COMC is a clinician completed clinical assessment of the subject's ability to communicate her choices or preferences, which can include the use of nonverbal means such as eye contact or gestures. The assessment is made on an 8-point Likert scale (0-7) with 0 denoting normal functioning and 7 the most severe impairment.
Time Frame: 40 Weeks Treatment Duration
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
score on a scale | -0.4 (0.13)

13. Secondary Outcome: Rett Syndrome Clinician Rating of Verbal Communication (RTT-VCOM) Change From Baseline to Week 40
Description: The RTT-VCOM is a clinician completed clinical assessment of the subject's ability to communicate verbally. The assessment is made on an 8-point Likert scale (0-7) with 0 denoting normal functioning and 7 the most severe impairment.
Time Frame: 40 Weeks Treatment Duration
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
score on a scale | -0.2 (0.07)

14. Secondary Outcome: Change From Baseline to Week 40 in Clinical Global Impression-Severity (CGI-S)
Description: The CGI-S is a 7-point scale that requires the clinician to rate the severity of the subject's illness at the time of assessment, relative to the clinician's experience with subjects who have the same diagnosis. Considering total clinical experience, a subject is assessed on severity of illness at the time of rating: 1=normal, not at all ill; 2=borderline ill; 3=mildly ill; 4= moderately ill; 5=markedly ill; 6=severely ill; or 7=extremely ill. Higher CGI-S scores denote more severe illness and less improvement in the illness.
Time Frame: 40 Weeks Treatment Duration
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
score on a scale | -0.1 (0.04)

15. Secondary Outcome: Rett Syndrome Caregiver Burden Inventory (RTT-CBI) Total Score (Items 1-24) Change From Baseline to Week 40
Description: The RTT-CBI consists of 24 negatively worded items (Items 1 through 24). Frequency ratings are on a 5-point Likert scale including: 0-never; 1-rarely; 2-sometimes; 3-frequently and 4-nearly always. The RTT-CBI also includes 2 positively worded items (items 25 and 26) that comprise the Optimism Index; this index will not be used for analysis. The total score ranging from 0 to 96 is calculated as the sum of the scores for Items 1-24.Higher scores signify higher caregiver burden.
Time Frame: 40 Weeks Treatment Duration
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
score on a scale | -1.9 (1.05)

16. Secondary Outcome: Impact of Childhood Neurologic Disability Scale (ICND) Total Score Change From Baseline to Week 40
Description: The ICND scale evaluates the effect of 4 health problems on 11 aspects of the child's or the family's life scored 0 ("Not at all"), 1 ("A little"), 2 ("Some"), 3 ("A lot"), or "Does not apply". The 4 health problems are 1) inattentiveness, impulsivity, or mood, 2) ability to think and remember, 3) neurologic or physical limitations, and 4) epilepsy. For each health problem, the score is calculated as the sum of the item scores. The ICND total score will be calculated as the sum of the average of each problem score multiplied by 11. The ICND total score ranges from 0 to 132. Higher ICND total scores indicate worse health problems. The ICND total score does not include the Overall Quality of Life Rating.
Time Frame: 40 Weeks Treatment Duration
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Trofinetide
Number analyzed (Participants) | 154
score on a scale | -5.8 (3.91)

ADVERSE EVENTS:
Time Frame: 44 weeks (including 40-week open-label treatment period and 30-day safety follow-up period)
Arm/Group | Trofinetide
All-Cause Mortality (participants affected / at risk) | 0/154
Serious Adverse Events (participants affected / at risk) | 19/154
Other Adverse Events (participants affected / at risk) | 114/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trofinetide (N=154)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Pneumonia (Infections and infestations) | 4 (6)
Rhinovirus infection (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Enterovirus infection (Infections and infestations) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Peritoneal abscess (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1)
Vaginal abscess (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Seizure (Nervous system disorders) | 5 (6)
Status epilepticus (Nervous system disorders) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trofinetide (N=154)
Diarrhoea (Gastrointestinal disorders) | 91 (129)
Vomiting (Gastrointestinal disorders) | 39 (58)
Pyrexia (General disorders) | 11 (14)
COVID-19 (Infections and infestations) | 16 (16)
Upper respiratory tract infection (Infections and infestations) | 12 (14)
Urinary tract infection (Infections and infestations) | 9 (14)
Weight decreased (Investigations) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 10 (11)
Seizure (Nervous system disorders) | 10 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT04279314/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT04279314/SAP_001.pdf